CLINICAL TRIAL: NCT03578120
Title: Immunising Mums Against Pertussis 3
Acronym: iMAP3
Status: Completed | Type: Observational
Sponsor: St George's, University of London (Other)
Collaborators: University of Oxford (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 17.0269
Record Dates: First submitted 2018-04-19; First posted 2018-07-05 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Whooping Cough; Maternal Vaccine Exposure; Immunization; Infection
MeSH Terms: conditions — Whooping Cough; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood sample to access serum sample to investigate antibody response towards pre-school booster vaccination
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- iMAP2 participants where their mothers received REPEVAX: Children who participated in iMAP2 study whose mothers received a pertussis-containing vaccine during pregnancy called REPEVAX
  Interventions: Biological: Pre-school booster vaccine
- iMAP2 participants where their mothers received BOOSTRIX-IPV: Children who participated in iMAP2 study whose mothers receives a pertussis-containing vaccine during pregnancy called BOOSTRIX-IPV
  Interventions: Biological: Pre-school booster vaccine
- iMAP2 participants where their mothers received no vaccine: Children who participated in iMAP2 study whose mothers did not receive a pertussis-containing vaccine during pregnancy
  Interventions: Biological: Pre-school booster vaccine

INTERVENTIONS:
Biological: Pre-school booster vaccine — Routine vaccination with pre-school booster vaccine

SUMMARY:
This study will aim to recruit at least 70 children who participated in the iMAP2 study whose mothers received a pertussis vaccine in pregnancy as part of the iMAP2 trial and at least 15 children born to mothers who did not receive a pertussis vaccine in pregnancy. Blood samples will be obtained prior to and one month after the routine preschool booster vaccination and vaccine responses compared between children whose mothers received one of two pertussis vaccines or no pertussis vaccine in pregnancy. Children will be vaccinated with the routine booster vaccines by the study team on the same visit as the pre-vaccination bloods are taken.

DETAILED DESCRIPTION:
In the UK, all pregnant women are offered a whooping cough-containing vaccine during pregnancy. This protects newborn infants against whooping cough, but there have been some concerns that this vaccination in pregnancy may affect the response to childhood vaccinations.

A preceding study called immunising Mums Against Pertussis 2 (iMAP2) was conducted involving pregnant women randomised to receive one of two different whooping cough-containing vaccines, with a control group also recruited, and the antibody levels in their infants were measured at age 2, 5 and 13 months.

This study, immunising Mums Against Pertussis 3 (iMAP3), is a follow up study of children who participated in iMAP2, to investigate the sustained impact of whooping cough vaccination in pregnancy on childhood vaccine responses.

This study will investigate the antibody levels in these children before and after the routine pre-school booster (DTaP/IPV vaccination) vaccine. It will help the Department of Health continue to ensure the best protection is offered to the population.

Those eligible for the study are children who participated in the iMAP2 study who have reached the age for pre-school booster vaccination (from age 3 years 4 months).

The study period will be approximately 4-6 weeks with two study visits. The first visit will take place when the child is around 3 years and 4 months of age. After informed consent a blood sample will be obtained followed by administration of the pre-school booster vaccine. At the second visit another blood sample will be obtained. These blood tests will measure the level of protective antibody against the components of the pre-school booster vaccine. Visits will take place either in the child's home or at a suitable clinical setting within the study team's sites.

The study will be run by St. George's, University of London, in collaboration with St George's University Hospitals NHS Foundation Trust, Oxford Vaccine Group and Bristol Children's Vaccine Centre.

ELIGIBILITY:
Inclusion Criteria:

* Age eligible for routine pre-school booster vaccinations (i.e. from 3 years and 4 months of age)
* Participated in the iMAP2 trial
* Informed consent by a parent or legal guardian

Exclusion Criteria:

* Permanent exclusion criteria:

  * Fulfil any of the contraindications to vaccination specified in The Green Book on Immunisation (https://www.gov.uk/government/organisations/public-health-england/series/immunisation-against-infectious-disease-the-green-book)
  * Received any additional pertussis containing vaccine after the routine 16 week booster
  * Previous or concurrent participation in an interventional study other than iMAP2 if, in the opinion of the investigator, this may influence the objectives of this study
* Temporary exclusion criteria:

  * If the child has an axillary/aural temperature ≥ 38°C then vaccination and blood sampling will be postponed until resolution of fever. If the child is acutely unwell, vaccination will be postponed until resolution
  * If the child is receiving antibiotics (other than long term prophylaxis) vaccination should be postponed until 48 hours after the conclusion of the course

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children who participated in the iMAP2 study of age to receive the routine pre-school booster vaccinations (i.e. from 3 years and 4 months of age)
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Fold-difference in anti-PT IgG geometric mean concentration (GMC) in children prior to booster vaccination | Up to a maximum of 3 years from the date of the last recruited participant
  To compare anti-pertussis toxin (PT) IgG concentrations at preschool age (around 3 years 4 months) and before receipt of the routine pre-school booster vaccine, in children born to mothers who received REPEVAX, BOOSTRIX-IPV or no pertussis containing vaccine in pregnancy.

SECONDARY OUTCOMES:
Fold-difference in anti-PT IgG geometric mean concentration (GMC) in children one month after booster vaccination | Up to a maximum of 3 years from the date of the last recruited participant
  To compare anti-pertussis toxin (PT) IgG concentrations at one month after receipt of the pre-school booster vaccine in children born to mothers who received REPEVAX, BOOSTRIX-IPV or no pertussis containing vaccine in pregnancy.
GMC of IgG to pertussis antigens (PT, PRN, FHA and FIM 2 and 3) prior to and one month after booster vaccination | Up to a maximum of 3 years from the date of the last recruited participant
  To compare antibody concentrations to other pertussis antigens [IgG to filamentous haemagglutinin (FHA) and fimbrial antigens 2 and 3 (FIM 2 and 3)], before and one month after receipt of a pre-school booster vaccine in children born to mothers who received REPEVAX, BOOSTRIX-IPV or no pertussis containing vaccine in pregnancy.
Anti-tetanus toxoid IgG GMC and anti-diphtheria toxoid IgG GMC prior to and one month after booster vaccination | Up to a maximum of 3 years from the date of the last recruited participant
  To compare antibody concentrations / titres to tetanus toxoid and diphtheria toxoid before and one month after receipt of a pre-school vaccine in children born to mothers who received REPEVAX, BOOSTRIX-IPV or no pertussis containing vaccine in pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Paul T Heath, MBBS FRCPCH, Principal Investigator — St George's, University of London
Locations (3):
- United Kingdom (3):
  - Gloucestershire NHS Trust, Gloucester
  - St George's, University of London, London
  - Oxford Vaccine Group, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sapuan S, Andrews N, Hallis B, Hole L, Jones CE, Matheson M, Miller E, Snape MD, Heath PT. An observational, cohort, multi-centre, open label phase IV extension study comparing preschool DTAP-IPV booster vaccine responses in children whose mothers were randomised to one of two pertussis-containing vaccines or received no pertussis-containing vaccine in pregnancy in England. Vaccine. 2022 Nov 22;40(49):7050-7056. doi: 10.1016/j.vaccine.2022.10.005. Epub 2022 Oct 20. PMID 36272877